CLINICAL TRIAL: NCT06162624
Title: Pilot Effectiveness Trial of an ACT Self-help Workbook Tailored Specifically for Prisons
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-1590; 1R34MH132663-01A1 (NIH); Protocol Version 07/02/25 (Other: UW Madison); A538900 (Other: UW Madison); SMPH/PSYCHIATRY/PSYCHIATRY (Other: UW Madison)
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Anxiety; Depression; Depression, Anxiety; Anxiety Disorders
Keywords: incarcerated
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Acceptance and Commitment Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT workbook (Experimental)
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Control workbook (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — ACT: Therapy that builds in traditional cognitive behavioral therapy principles but emphasizes different processes in behavior change. Delivered over 8 weeks of self-guided study and homework assignments.
  Arms: ACT workbook
Behavioral: Cognitive Behavioral Therapy (CBT) — As control condition, reflective journaling will be used.
  Arms: Control workbook

SUMMARY:
The goal of this research study is to adapt an ACT-self-help workbook to the prison setting and determine the feasibility acceptability, and effectiveness of this workbook.

Participants can expect to be in the study for 13 weeks.

DETAILED DESCRIPTION:
The Specific Aims of the proposed study correspond directly to the three-step process.

1. In Step 1 (Specific Aim #1), identify the necessary adaptations to the content, language, and format of an ACT-based self-help workbook through stakeholder input.
2. In Step 2 (Specific Aim #2), refine the workbook and its delivery based on feedback from incarcerated individuals who complete the workbook.
3. In Step 3 (Specific Aim #3), determine the feasibility, acceptability and preliminary effectiveness of the ACT self-help workbook in a prison setting. Primary clinical outcome measure will be depression, secondary clinical outcome measure will be anxiety.

For each participant assigned to a condition, a study team member will meet with them individually to provide them with a copy of the workbook. During this meeting, the study team member will inform the participant that they should complete one chapter per week.

Participants will complete a Pre-Treatment Assessment prior to distribution of the workbook; a Mid-Treatment Assessment four weeks after the distribution of the workbook; a Post-Treatment Assessment #1 eight weeks after distribution of the workbook (when the workbook should be completed); Focus group (after completion of workbook) and, a Post-Treatment Assessment #2 twelve weeks after distribution of the workbook.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Reading level of 6th grade or higher determined by the Wide Range Achievement Test
* Moderate or severe anxiety and/or depression determined by the Beck Depression Inventory-II (BDI-II) and Beck Anxiety Inventory (BAI)
* No active self-harm or active suicidal intent
* No scheduled transfer or release for at least three months
* Must be willing and able to participate, including having permission and ability to use study materials, such as paper and a writing utensil

Exclusion Criteria:

* Unable to provide informed consent
* Active self-harm or suicidal intent
* Scheduled transfer or release within three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Eligible participants | Study duration, up to 1 year
  Feasibility will be assessed by measuring eligibility - percentage of individuals who meet inclusion criteria versus percentage of individuals who are excluded.
Participants who choose to participate | Study duration, up to 1 year
  Feasibility will be assessed by measuring the percentage of eligible individuals who choose to participate in the study.
Percentage of participants that complete all 8 weeks | Study duration, up to 1 year
  Feasibility will be assessed by measuring the percentage of participants who complete all treatment activities
Qualitative Summary of Reasons for Attrition | Study duration, up to 1 year
  Feasibility will be assessed qualitatively by asking participants who leave the study, why they decided to stop. Responses will be coded for themes and summarized with participant counts.
Number of Participants referred for Follow up care | Up to 13 weeks
  Safety will be measured through participant self-report suicidal or self-harm ideation, using the Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS is a questionnaire designed to assess the level of risk for self-harm. Any participant that indicates active suicidal ideation with intent to act or active suicidal ideation with a specific plan on the C-SSRS will be referred for follow up care.
Participant Satisfaction | Up to 13 weeks
  Acceptability of the method will be assessed through Client Satisfaction Questionnaire (CSQ-8), which is an 8 item survey with potential scores of 8-32 with higher scores indicating greater satisfaction.
Change in Mental Health: Flexibility | Baseline to 13 weeks
  The Multidimensional Psychological Flexibility Inventory (MPFI) assesses the 12 dimensions of flexibility and inflexibility. Responses have point values from 1 to 6, where higher scores reflect higher levels of the dimension being assessed by each set of items.
Change in Mental Health: Automatic Thoughts | Baseline to 13 weeks
  The Automatic Thoughts Questionnaire lists are a variety of thoughts that pop into people's heads. Participants read each thought and indicate how frequently, if at all, the thought has occurred over the past week. 30 questions with a scale of 1-5, with 1 = not at all and 5 = all of the time. Higher scores indicate higher frequency of automatic thoughts.
Change in BAI Score | Baseline to 13 weeks
  Beck Anxiety Inventory (BAI) is a 21-item self-reported questionnaire which measures the existence and severity of symptoms of anxiety. Each of the 21 items on BAI tool represents an anxiety symptom. A total score of 0 - 7 is interpreted as a "Minimal" level of anxiety; 8 - 15 as "Mild"; 16 - 25 as "Moderate", and 26 - 63 as "Severe".
Change BDI-II Score | Baseline to 13 weeks
  Beck Depression Inventory (BDI-II) Scale is a 21-item self-reported questionnaire which measures the existence and severity of symptoms of depression. Each of the 21 items on BDI-II tool represents a depressive symptom. The symptoms are each scored on a 4-point Likert scale of 0 to 3 (0=symptom is absent; 3=symptom is severe). Scores for each symptom are added up to obtain the total scores for all 21 items. Total score ranges from 0-63; of which 0-8 is considered no depression, 0-13 is minimal depression, 14-19 is mild depression, 20-28 is moderate depression and 29-63 is severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Koenigs, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No